CLINICAL TRIAL: NCT04808687
Title: Phase II Single-arm Trial of Nab-Paclitaxel and S-1 as Neoadjuvant Treatment of Patients With Resectable Pancreatic Cancer
Brief Title: Neoadjuvant Nab-Paclitaxel and S-1 in Resectable Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TZ-PC02
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Taxes; S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nab-paclitaxel and S-1 (Experimental): neoadjuvant chemotherapy with Nab-paclitaxel and S-1, repeat every 21 days for 2-4 cycles
  Interventions: Drug: Nab paclitaxel and S-1

INTERVENTIONS:
Drug: Nab paclitaxel and S-1 — Nab-Paclitaxel: 125 mg/m2 d1, 8, during each 3-week cycle. S-1: Body surface area < 1.25 m2, 40 mg bid; Body surface area ≥ 1.25 m2 < 1.50 m2, 50 mg bid; Body surface area ≥1.5 m2, 60 mg bid, d1-14;during each 3-week cycle.

SUMMARY:
There were limited data for nab-paclitaxel and S-1 in pancreatic cancer. To explore the efficacy and safety of neoadjuvant nab-paclitaxel combined with S-1 in patients with resectable pancreatic cancer (stage II and partial stage III defined according to the National Comprehensive Cancer Network definitions ), we designed this study. This study was a single-arm single center prospective phase II clinical study. A total of 72 subjects who meet the criteria will receive neoadjuvant chemotherapy of nab-paclitaxel and S-1 prior to pancreatectomy. Response was reported according to the Response Evaluation Criteria in Solid Tumors guidelines (RECIST, version 1.1) .The primary endpoint is objective response rate. The secondary endpoints include R0/R1 resection rate, disease free survival, overall survival and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed-consent form;
2. Treatment-naive PDAC with histological or cytological diagnosis;
3. Resectable pancreatic cancer stage II and partial stage III defined according to the National Comprehensive Cancer Network definitions;
4. Age≥18 years old and ≤70 years old;
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
6. BMI≥18.5 and NRS2002score<3;
7. Expected survival over 3 months;
8. Spared organ function satisfying the following laboratory data:leucocyte≥3.0x109/L,neutrophils≥1.5x109/L, hemoglobin≥ 9g/dL, platelets ≥100x109/L, total bilirubin ≤ 1.5 ULN; AST and ALT≤ 2.5 ULN; serum creatinine≤1.5ULN; PT and INR≤ 2.5 ULN;

Exclusion Criteria:

1. Severe Impaired organ functions;
2. Patients who had surgeries, chemotherapy or other treatments before inclusion;
3. Pregnant women or lactating women;
4. Ineligible by the discretion of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first,assessed up to 24 months
  Percentage of patients who achieve partial response (PR) or complete response(CR) based on Response Evaluation Criteria In Solid Tumors (RECIST1.1)

SECONDARY OUTCOMES:
R0/R1 resection rate | 2 years
  proportion of patients who achieved R0/R1 resection
Disease free survival | From date of randomization until the date of first documented progression or metastasis, assessed up to 12 months
  The time between operation and the relapse or metastasis of tumors or death
Overall survival | From date of randomization until the date of death from any cause or censored at the last day that the patient is documented to be alive, whichever came first, assessed up to 24 months
  The time between randomization and death from any cause or lost to follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No